CLINICAL TRIAL: NCT06893809
Title: Effects of Different Routes of Local Anesthetic Administration in Epidural Anesthesia for Transurethral Resection of The Prostate
Brief Title: Epidural Anesthesia for Transurethral Resection of The Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANEAH2010; Corresponding Author (Other: Başakşehir Cam and Sakura City Hospital)
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Epidural Catheter; Epidural Analgesia; Geriatric Cardiology; Urologic Disorders; Hemodynamic (MAP) Stability; Pain Management
Keywords: Transurethral resection of the prostate; epidural anesthesia
MeSH Terms: conditions — Urologic Diseases; Agnosia | interventions — Needles; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group N (Active Comparator): Group N (Needle)
  Interventions: Procedure: Epidural injection via catheter; Procedure: Combined epidural injection (needle and catheter)
- Group C (Active Comparator): Group C (Catheter)
  Interventions: Procedure: Epidural injection via Tuohy needle; Procedure: Combined epidural injection (needle and catheter)
- Group N/C (Active Comparator): Group N/C (Needle/Catheter)
  Interventions: Procedure: Epidural injection via Tuohy needle; Procedure: Epidural injection via catheter

INTERVENTIONS:
Procedure: Epidural injection via Tuohy needle — Local anesthetic was administered entirely through the Tuohy needle.
  Other Names: Epidural anesthesia - needle route
  Arms: Group C; Group N/C
Procedure: Epidural injection via catheter — Local anesthetic was administered entirely through the epidural catheter.
  Other Names: Epidural anesthesia - catheter route
  Arms: Group N; Group N/C
Procedure: Combined epidural injection (needle and catheter) — Half of the total local anesthetic dose was administered through the needle and half through the catheter.
  Other Names: Epidural anesthesia - combined route
  Arms: Group C; Group N

SUMMARY:
The aim of this study is to assess the effects of different routes of local anesthetic administration in epidural anesthesia applied to patients undergoing transurethral resection of the prostate (TUR-P). ASA I-III 60 patients were enrolled in the study. Patients were randomized into the following three groups: in Group N (needle), total dose of local anesthetic was administered through the Tuohy needle (n=20), in Group C (catheter), local anesthetic was administered through the epidural catheter (n=20) and in Group N/C (needle/catheter), local anestetic was administered half volume through the needle and half through the catheter (n=20). Hemodynamics, times to reach sensory block T10 (block levels), side effects, patient and surgeon satisfaction were evaluated.

DETAILED DESCRIPTION:
In urological procedures, the preferred anaesthetic modalities may be topical, regional or general. The decision is made by the anaesthesiologists based on patient age, sex, general condition and the surgical procedure to be performed. Transurethral procedures are frequently applied to geriatric patients, who are more likely to have comorbidities. In such cases, epidural anaesthesia may be preferred for geriatric patients.

In this study, we utilised various routes for the administration of local anaesthetics to induce epidural anaesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) due to benign prostatic hyperplasia. The study encompassed the evaluation of haemodynamic stability, the time to reach sensory block T10, the occurrence of side effects, and the levels of patient and surgeon satisfaction.

Following the approval of the hospital ethics committee, 60 male patients aged 40-75, ASA class I-III, scheduled for elective TUR-P surgery were enrolled in the study.According to the method of local anaesthetic administration, patients were randomly divided into three groups:

Group N (needle); total local anaesthetic administered through the Tuohy needle,Group C (catheter); local anaesthetic administered through the epidural catheter,Group NC (needle/catheter); 50% of local anaesthetic administered through the needle and 50% through the catheter.Patients underwent standard monitorisation in the operating theatre. Each patient received 0.03 mg/kg of midazolam intravenously following catheterisation with a 20-gauge intravenous cannula.Prior to the commencement of epidural block, patients were preloaded with 10 ml/kg of 0.9% isotonic saline infused over a 30-minute period. The hemodynamic parameters were then recorded before and after the premedication, following the epidural block, and every 5 minutes until the patient's sensory block level regressed to L1 dermatome.The epidural anaesthesia was then attempted with an 18-gauge Tuohy needle at the L3-4 interspinal level using the loss of resistance technique following infiltration with 2% lidocaine. Patients in Group N received a mixture of 8ml 2% prilocaine, 7ml 0.5% levobupivacaine and 50μg fentanyl through the epidural space using a Tuohy needle. Patients in Group C received the same drug combination through the epidural catheter. Patients in Group NC received half of the same drug combination through the needle and half through the epidural catheter. Patients were positioned in the right lateral decubitus position with thighs flexed up and neck flexed forward (fetal position), and then placed supine following drug administration.In all groups, time "0" was considered as the time that drug administration was started.

The sensory and motor block levels, heart rates and mean arterial blood pressure values, times to reach sensory block level T10, and side effects were recorded for all patients. Patient and surgeon satisfaction levels were evaluated using a 3-point satisfaction scale by an observer unaware of the study's objectives.Surgeon satisfaction was evaluated during the operation, and patient satisfaction was assessed in the recovery room before patients were transferred to their service bed.

Post-operatively, patients were admitted to the recovery room, the epidural catheter was removed following regression of sensory block to T10 dermatome, and patients were transferred to the service.

ELIGIBILITY:
Inclusion Criteria:

* Male undergoing transurethral prostatic resection,
* 40 to 75 years old,
* ASA-I-III
* Not using anticoagulants or antiaggregants,
* No peripheral neuropathy or muscle disease,
* Can be orientated and co-operated,
* No vertebral deformity,
* Body Mass Index <30,
* Patients consenting to epidural anaesthesia.

Exclusion Criteria:

* TUR-P operation will not be male,
* Female patients,
* ASA-IV,
* Not in the appropriate age range (40-75),
* Taking anticoagulants or antiaggregants, Previous lumbar surgery or skeletal deformity in the lumbar region,
* Peripheral neuropathy, neuromuscular or neuropsychiatric disease,
* Alcohol or drug addiction,
* Obese with a body mass index >30,
* History of frequent analgesic use,
* Patients shorter than 155 cm and taller than 180 cm,
* Who refused epidural anaesthesia,
* Patients without orientation and co-operation.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients undergoing transurethral prostatic resection
Enrollment: 60 (Actual)
Dates: Start 2010-01-02 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NERMİN GÖĞÜŞ, Prof.Dr., Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Numune Education and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All results
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Timeless
Access Criteria: All researchers can access all information.
URL: https://www.jscimedcentral.com/public/assets/articles/anesthesiology-4-1050.pdf

REFERENCES:
- [Background] Barbosa FT, Castro AA. Neuraxial anesthesia versus general anesthesia for urological surgery: systematic review. Sao Paulo Med J. 2013;131(3):179-86. doi: 10.1590/1516-3180.2013.1313535. PMID 23903267
- [Background] Kim JH, Lee JS, Kim DY. Direction of catheter insertion and the incidence of paresthesia during continuous epidural anesthesia in the elderly patients. Korean J Anesthesiol. 2013 May;64(5):443-7. doi: 10.4097/kjae.2013.64.5.443. Epub 2013 May 24. PMID 23741568
- [Background] Horlocker TT, Abel MD, Messick JM Jr, Schroeder DR. Small risk of serious neurologic complications related to lumbar epidural catheter placement in anesthetized patients. Anesth Analg. 2003 Jun;96(6):1547-1552. doi: 10.1213/01.ANE.0000057600.31380.75. PMID 12760972
- [Background] Yun MJ, Kim YC, Lim YJ, Choi GH, Ha M, Lee JY, Ham BM. The differential flow of epidural local anaesthetic via needle or catheter: a prospective randomized double-blind study. Anaesth Intensive Care. 2004 Jun;32(3):377-82. doi: 10.1177/0310057X0403200313. PMID 15264734
- [Background] Omote K, Namiki A, Iwasaki H. Epidural administration and analgesic spread: comparison of injection with catheters and needles. J Anesth. 1992 Jul;6(3):289-93. doi: 10.1007/s0054020060289. PMID 15278539
- [Background] Crochetiere CT, Trepanier CA, Cote JJ. Epidural anaesthesia for caesarean section: comparison of two injection techniques. Can J Anaesth. 1989 Mar;36(2):133-6. doi: 10.1007/BF03011434. PMID 2650896
- [Background] Visser WA, Lee RA, Gielen MJ. Factors affecting the distribution of neural blockade by local anesthetics in epidural anesthesia and a comparison of lumbar versus thoracic epidural anesthesia. Anesth Analg. 2008 Aug;107(2):708-21. doi: 10.1213/ane.0b013e31817e7065. PMID 18633056
- [Background] Cesur M, Alici HA, Erdem AF, Silbir F, Yuksek MS. Administration of local anesthetic through the epidural needle before catheter insertion improves the quality of anesthesia and reduces catheter-related complications. Anesth Analg. 2005 Nov;101(5):1501-1505. doi: 10.1213/01.ANE.0000181005.50958.1E. PMID 16244020
- [Background] Ulker B, Erbay RH, Serin S, Sungurtekin H. Comparison of spinal, low-dose spinal and epidural anesthesia with ropivacaine plus fentanyl for transurethral surgical procedures. Kaohsiung J Med Sci. 2010 Apr;26(4):167-74. doi: 10.1016/S1607-551X(10)70025-5. PMID 20434097
- [Background] Sorenson RM, Pace NL. Anesthetic techniques during surgical repair of femoral neck fractures. A meta-analysis. Anesthesiology. 1992 Dec;77(6):1095-104. doi: 10.1097/00000542-199212000-00009. PMID 1466461
- [Background] Bernstein S, Malhotra V. Regional anesthesia for genitourinary surgery. In Malhotra V (ed): Anesthesia for Renal And Genitourinary
- [Background] Blake DW. The general versus regional anaesthesia debate: time to re-examine the goals. Aust N Z J Surg. 1995 Jan;65(1):51-6. doi: 10.1111/j.1445-2197.1995.tb01748.x. PMID 7818424
- [Background] Morgan GE, Mikhail MS, Murray MJ, Larson CP. Regional Anesthesia &Pain Management, Clinical Anesthesiology. 3rd edition. Los Angeles:
- [Background] Tsui BC, Wagner A, Finucane B. Regional anaesthesia in the elderly: a clinical guide. Drugs Aging. 2004;21(14):895-910. doi: 10.2165/00002512-200421140-00001. PMID 15554749
- See also: jscimedcentral — https://www.jscimedcentral.com/public/assets/articles/anesthesiology-4-1050.pdf
- Available data/document: Clinical Study Report: https://www.jscimedcentral.com — https://www.jscimedcentral.com/public/assets/articles/anesthesiology-4-1050.pdf — Int J Clin Anesthesiol 4(1): 1050 (2016)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 2010 study at Ankara Numune Education and Training Hospital examined patients 40-75 undergoing transurethral prostatectomy. Excluded were those with certain health issues or specific procedures. Patients gave consent before being divided into three groups: NC for needle and catheter; C for catheter only; N for needle only.
Pre-assignment Details: Patients above ASA-III, with peripheral neuropathy, neuromuscular or neuropsychiatric disease, alcohol or drug addiction, obese (body mass index >30), history of hypersensitivity to local anesthetic agents, scoliosis, low back pain or history of lumbar surgery, bleeding, coagulation disorder, infection, history of frequent analgesic use, shorter than 155 cm and taller than 180 cm were excluded from the study.
Groups:
- Group N: Group N (Needle)
  The group in which the dose of local anaesthetic to be used for epidural anaesthesia is administered exclusively through the needle.
- Group C: Group C (Catheter)
  The group is characterised by the administration of the local anaesthetic dose for epidural anaesthesia, which is administered exclusively through the epidural catheter.
- Group N/C: Group N/C (Needle/Catheter)
  The total dose of local anaesthetic administered for epidural anaesthesia was divided into two equal parts; the first part was injected through the touhy needle, and the second part was administered after the epidural catheter had been inserted.
Period: Overall Study
Arm/Group | Group N | Group C | Group N/C
Started | 20 (In Group N, after standard monitoring and sedation, the local anesthetic mixture was injected directly into the epidural space through the needle, the catheter was advanced 2-3 cm in the epidural space in a cranial direction. The catheter was appropriately fixed to the skin.) | 20 (After identifying the epidural space, a 22-gauge Touhy needle was used to advance the catheter 2-3 cm in the epidural space cranially. The needle was then withdrawn, and the catheter was fixed to the skin. The same dose of local anesthetic mixture used in the needle group was injected into the epidural space in this group.) | 20 (Group N/C participants underwent intravenous access with a 20-gauge cannula on the back of the hand after standard monitoring in the operating room, followed by epidural block and sedation. Half the local anesthetic mixture was injected through the Touhy needle after its epidural space was identified, while the other half was injected via the catheter.)
Completed | 20 (The study concluded upon reaching the predetermined number of patients.) | 20 (The study concluded upon reaching the predetermined number of patients.) | 20 (The study concluded upon reaching the predetermined number of patients.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group N (Needle): In this study, we utilised various routes for the administration of local anaesthetic, with the objective of achieving epidural anaesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) for benign prostatic hyperplasia. The study encompassed the evaluation of haemodynamic stability, the times to reach T10 sensory block, the occurrence of side effects, and the levels of patient and surgeon satisfaction. Following approval by the hospital ethics committee, a total of 60 male patients aged between 40 and 75 years, with an American Society of Anesthesiologists (ASA) classification of I-III, scheduled for elective transurethral prostate surgery (TUR-P), were included in the study. Patients were randomly divided into three groups according to the type of local anaesthetic administration: Group N (needle); the total local anaesthetic dose was administered through a Tuohy needle.
- Group C (Catheter): In this study, we used various routes for local anaesthetic administration to achieve epidural anaesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) for benign prostatic hyperplasia. The study included evaluation of haemodynamic stability, times to reach T10 sensory block, occurrence of side effects and patient and surgeon satisfaction levels. Following approval by the hospital ethics committee, a total of 60 male patients aged 40-75 years, American Society of Anaesthesiologists (ASA) classification I-III, scheduled for elective transurethral prostate surgery (TUR-P) were included in the study. Patients were randomly divided into three groups according to the type of local anaesthetic administration: Group C (Catheter); the total dose of local anaesthetic was administered through an epidural catheter.
- Group N/C (Needle/Catheter): In this study, we used various routes for local anaesthetic administration to achieve epidural anaesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) for benign prostatic hyperplasia. Haemodynamic stability, times to reach T10 sensory block, occurrence of side effects and patient and surgeon satisfaction levels were evaluated. Following approval of the hospital ethics committee, a total of 60 male patients aged 40-75 years, American Society of Anaesthesiologists (ASA) classification I-III, scheduled for elective transurethral prostate surgery (TUR-P) were included in the study. The patients were randomly divided into three groups according to the type of local anaesthetic administration: In group N/C (Needle/Catheter), half of the total local anaesthetic dose was administered through touhy needle and the remaining half through epidural catheter.
- Total: Total of all reporting groups
Arm/Group | Group N (Needle) | Group C (Catheter) | Group N/C (Needle/Catheter) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 20 | 20 | 20 | 60
Age [Mean (Standard Deviation); unit: years] | 65.45 (8.56) | 61.05 (9.71) | 64.20 (7.01) | 63.57 (8.56)

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Sensory Block at T10
Description: Times to reach sensory block T10 (block levels)
Time Frame: Within 20 minutes after anesthetic administration
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Group N: Group N (Needle)
  Grup C: Local anesthetic was administered through the epidural catheter.
  Grup N/C: (needle/catheter); half of the local anesthetic was administered through the needle and half through the catheter.
- Group C: Group C (Catheter)
  Grup N: In this study, we used different paths to administer local anesthetic to achieve epidural anesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) due to benign prostatic hyperplasia and evaluated hemodynamic stability, times to reach sensory block T10, side effects as well as patient and surgeon satisfaction. After the approval of the hospital ethics committee, 60 male patients aged 40-75, ASA class I-III scheduled for elective TUR-P surgery were enrolled in the study. According to the path of local anesthetic administration, patients were randomly divided into three groups:
  Group N (needle); total local anesthetic dose was administered through the Tuohy needle.
  Grup N/C: (needle/catheter); half of the local anesthetic was administered through the needle and half through the catheter.
- Group N/C: Group N/C (Needle/Catheter)
  Grup N: In this study, we used different paths to administer local anesthetic to achieve epidural anesthesia in patients scheduled for transurethral resection of the prostate (TUR-P) due to benign prostatic hyperplasia and evaluated hemodynamic stability, times to reach sensory block T10, side effects as well as patient and surgeon satisfaction. After the approval of the hospital ethics committee, 60 male patients aged 40-75, ASA class I-III scheduled for elective TUR-P surgery were enrolled in the study. According to the path of local anesthetic administration, patients were randomly divided into three groups:
  Group N (needle); total local anesthetic dose was administered through the Tuohy needle.
  Grup C: Local anesthetic was administered through the epidural catheter.
Arm/Group | Group N | Group C | Group N/C
Number analyzed (Participants) | 20 | 20 | 20
Minutes | 15.25 (1.97) | 10.50 (1.54) | 11.25 (2.22)
Statistical Analysis 1: Comparison: Group N vs Group C vs Group N/C; Sixty male patients scheduled for TURP surgery were divided into three equal groups. The results were evaluated at a 95% confidence interval, with significance set at p < 0.05. This was achieved using SPSS 15.0. Between-group comparisons were performed using One-way ANOVA, Kruskal-Wallis, Wilcoxon Signed Ranks, and Friedman tests. Within-group comparisons used Wilcoxon Signed Ranks tests, and Friedman tests were used for differences over time; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Net) = 10, 95% CI 2-sided [10 to 20], Standard Deviation 5
Statistical Analysis 2: Comparison: Group N vs Group C vs Group N/C; The aim of this analysis is to compare the three groups in terms of patient and surgeon satisfaction using a superiority approach. The null hypothesis is that there is no difference in satisfaction scores between the groups. Statistical significance was set at p < 0.05; Test type: Superiority; p > 0.05, Kruskal-Wallis — No adjustment for multiple comparisons was applied. Non-parametric method used due to ordinal scale structure; Mean Difference (Final Values) = 0, 95% CI 2-sided [0 to 0], Standard Deviation 0 — Patient and surgeon satisfaction were compared across study arms

2. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in Systolic Blood Pressure from Sedation to 20 Minutes Post-Epidural Block
Time Frame: From 5 minutes after sedation to 20 minutes after epidural block
Population: All randomized participants (n=60), equally distributed into three groups (n=20 per group), completed the study and were included in the final analysis. No participants were withdrawn or excluded after randomization. The analysis was performed on a per-protocol basis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group N | Group C | Group N/C
Number analyzed (Participants) | 20 | 20 | 20
mmHg
  Sedation SBP (mean ± SD) | 126.70 (13.80) | 123.80 (8.61) | 126.70 (13.80)
  Post-Block 20th Min SBP (mean ± SD) | 116.80 (16.04) | 116.40 (11.99) | 121.10 (13.50)

3. Secondary Outcome: Maximum Sensory Block Level at the 20th Minute Post-Epidural Block
Description: Dermatomes were converted to numerical scores for statistical analysis:
  L1 = 1, T12 = 2, T10 = 3, T8 = 4, T6 = 5. Maximum sensory block level was assessed by converting dermatomal levels to numerical scores: L1 = 1, T12 = 2, T10 = 3, T8 = 4, T6 = 5. Higher scores indicate higher (more cephalad) dermatomal levels, which are considered better outcomes in terms of anesthetic spread.
Time Frame: 20 minutes after epidural administration
Measure: Mean (Standard Deviation); unit: Score on a 1-5 scale
Arm/Group | Group N | Group C | Group N/C
Number analyzed (Participants) | 20 | 20 | 20
Score on a 1-5 scale | 3.20 (0.52) | 4.10 (0.55) | 4.25 (0.54)
Statistical Analysis 1: Comparison: Group N vs Group C vs Group N/C; Test type: Superiority; p = 0.05, Kruskal-Wallis; Non-parametric test used due to ordinal scale and non-normal distribution; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [0.5 to 1.6] — Sensory block levels compared across study arms using numerical dermatomal codes

4. Secondary Outcome: Motor Block Intensity Based on Bromage Score at 20 Minutes
Description: Motor block was assessed using the modified Bromage scale:
  0 = No motor block
  1. = Partial block (able to move knees and feet)
  2. = Moderate block (unable to flex knees, able to move feet)
  3. = Complete block (unable to move feet or legs). Scores range from 0 (best outcome, least block) to 3 (worst outcome, complete motor block). Lower scores indicate better functional recovery.
Time Frame: 20 minutes after epidural block administration
Measure: Mean (Standard Deviation); unit: Score on a 0-3 scale
Arm/Group | Group N | Group C | Group N/C
Number analyzed (Participants) | 20 | 20 | 20
Score on a 0-3 scale | 0.30 (0.66) | 0.60 (1.00) | 0.20 (0.62)

5. Secondary Outcome: Degree of Sensory Block Regression at 60 Minutes Post-Epidural Block
Description: Sensory block regression at 60 minutes post-epidural block was assessed by converting dermatomal levels into numerical scores: L1 = 1, T12 = 2, T10 = 3. This scoring reflects the highest remaining level of sensory block at 60 minutes. Lower scores indicate greater regression of the block, meaning faster recovery. The minimum score is 1 and the maximum is 3.
Time Frame: 60 minutes after epidural block administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a 1-3 scale
Arm/Group | Group N | Group C | Group N/C
Number analyzed (Participants) | 20 | 20 | 20
Score on a 1-3 scale | 2.3 (0.47) | 2.8 (0.86) | 2.5 (0.61)
Statistical Analysis 1: Comparison: Group N vs Group C vs Group N/C; Test type: Superiority; p < 0.05, Kruskal-Wallis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.07 to 0.93], Standard Error of Mean 0.22 — Dermatomal regression levels were compared across groups at 60 minutes

ADVERSE EVENTS:
Time Frame: Eight months
Description: Allergy to drugs, Intravenous administration of drugs, Haemorrhage/bruising/hematoma/infection, Epidural haemorrhage , Puncturing the dura mater, Severe headaches, Blocking at high level, Haemodynamic instability, Cardiac and respiratory arrest, Total spinal nerve blockade following local anesthetic injection. SCTID: 405363008 Local anesthetic block inadequate. SCTID: 405364002
Arm/Group | Group N | Group C | Group N/C
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The study's findings are subject to at least two limitations. Firstly, the participants were members of an advanced age group, which is known to be associated with an increased prevalence of comorbidities. Secondly, the duration of surgery was longer than expected, which may be indicative of a more complex and time-consuming surgical procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2010-11-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT06893809/SAP_000.pdf